CLINICAL TRIAL: NCT01890668
Title: Efficacy Assessment of Early Osteopathic Manipulative Treatment (OMT) in the Management of Suboptimal Breastfeeding Behaviour in Healthy Newborns. A Prospective Monocentric Randomized Double-blinded Study.
Brief Title: Efficacy Assessment of Osteopathic Manipulative Treatment in the Suboptimal Breastfeeding Behaviour
Acronym: NEOSTEO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RC12_0379
Record Dates: First submitted 2013-06-21; First posted 2013-07-02 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: Breast Feeding, Exclusive
Keywords: Breastfeeding behaviour; OMT (Osteopathic Manipulative Treatment); suboptimal infant breastfeeding behaviour; healthy newborns
MeSH Terms: conditions — Breast Feeding | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Osteopathic Manipulative Treatment (Experimental): Randomization and first OMT will take place at discharge (Day 3); second osteopathic therapy will be performed by the same osteopath practitioner at Day10.
  Interventions: Other: Osteopathic Manipulative Treatment
- Control group (Placebo Comparator): Control group consists in classical medical and paramedical breastfeeding support. OMT on the newborn will be realized by osteopath dissimulated behind a screen. Placebo OMT consists to mimic, without the knowledge of parents, osteopathic techniques on a dolly.
  Interventions: Other: No Osteopathic manipulative Treatment

INTERVENTIONS:
Other: Osteopathic Manipulative Treatment — Visit 1 between H60 and discharge :
  Interview (pregnancy step, initiation of breastfeeding, baby posture…) Osteopathic Clinical exam (osteopathic specific diagnosis, mobility…) Osteopathic Manipulative Treatment by sweet osteopathic mobilization Time of intervention = 30 to 45 min Visit 2 : 7 days after visit 1 (+/- 24H) with the same procedure
  To keep the blinded procedure the interventions will be realized behind a screen, allowing interactions with parents but depriving their visibility.
  A telephone contact will be perform at M1 (one month of life) to assess breastfeeding persistence and collect questionnaire data.
  Two others telephone contacts will be perform at 3 months and 6 months to precise breastfeeding interruption date.
  The follow-up for each patient is 6 months
  Arms: Osteopathic Manipulative Treatment
Other: No Osteopathic manipulative Treatment — Visit 1 between H60 and discharge :
  Interview (pregnancy steps, initiation of breastfeeding, baby posture…) Osteopathic Clinical exam and Treatment will not be realized. Newborn will be undressed, lying naked (covered with polar sheet) on the exam table, dissimulated to parents by adequate screen. The osteopathic procedure will take place on a dolly to mimic from an indiscernible manner, osteopathic management.
  Time of intervention = 30 to 45 min Visit 2: 7 days after visit 1 (+/- 24H) with the same procedure.
  To keep the blinded procedure the interventions will be realized behind a screen, allowing interactions with parents but depriving their visibility.
  A telephone contact will be perform at M1 (one month of life) to assess breastfeeding persistence and collect questionnaire data.
  Two others telephone contacts will be perform at 3 months and 6 months to precise breastfeeding interruption date.
  The follow-up for each patient is 6 months
  Arms: Control group

SUMMARY:
Breastfeeding is one of the prime factors of long-term health protection in newborns, for nutritional, immunological and developmental reasons. In France there is a wide inter-regional variability of breastfeeding rates at discharge. This variability associates different factors involving both, mothers, birth conditions, newborns and mother-child couple. Some approaches, including osteopathy, aim to support early breastfeeding difficulties. As many others non-conventional medicines, there is a huge and growing interest for this alternative therapy and a spontaneous recourse in the first months of life. Nevertheless, neither efficacy nor the benefits have been studied. Thus, our objective is to evaluate for the first time in France, in a randomized, double-blinded design, the efficacy of early osteopathic manipulative treatment (OMT), in suboptimal breastfeeding behaviour healthy newborns.

128 couples mother-child will be randomized in two groups: with or without osteopathic intervention on the newborn.

ELIGIBILITY:
Inclusion Criteria:

* Healthy newborn ≥ 38 weeks of gestation,
* Suboptimal breastfeeding behavior defined by an IBFATmax score <10 after 2 assessments.(IBFATmax score = maximal score of Infant Breast Feeding Assessment Tool)
* And/ or presence of persistent severe pain (VAS> 5) at hospital discharge,
* And / or the presence of nipples cracks, grades 2-5 on the NTS scale
* Maternal Project of exclusive breastfeeding.
* Parental informed and consent form signed

Exclusion Criteria:

* Prematurity defined by a gestation <38 weeks
* Hypotrophy
* Maternal obesity (BMI>40)
* Multiple pregnancy
* Congenital malformation
* Neonatal pathology incompatible with efficient lactation initiation.
* Mothers minor or major and / or under guardianship and / or with poor understanding of French language
* Previous history of maternal breast surgery or umbilicated nipple
* IBFAT score max >10 on at least one of the two assessment at Day3.
* Medical contraindication to osteopathy: bone injury (fracture), tendon or ligament (sprain, dislocation etc ...) in the newborn incompatible with effective mobilization.
* Parental consent withdrawal.
* Neonatal pathology incompatible with breastfeeding follow-up in the first month of life.

Ages: 1 Day to 4 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 128 (Actual)
Dates: Start 2013-07; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Efficacy assessment of osteopathic treatment on breastfeeding failure at 1 month of life. | at 1 month of life.
  compare of breastfeeding failure percentage at one month of life between the two arms

SECONDARY OUTCOMES:
Compare IBFAT score (Infant Breast Feeding Assessment Tool score) | at 10 days of life
  compare the IBFAT score between the two consultation Cs1(day 3) and Cs2 (day 10)
Maternal satisfaction assessment | at one month of life
  assessment of maternal satisfaction between the Cs1, Cs2 and the visit at one month, by VAS
Safety assessment measured by per-treatment DAN score | at 3 days of life
Preventive efficacy of osteopathic treatment on nipple cracks, measured by the number of nipple cracks | at one month of life
Description of newborns behaviour during the first month of life (sleeping/awakening rhythm, cries and breastfeeding durations etc…) according treatment arm. | at one month of life
Description of breastfeeding initiation during the first month of life. | at one month of life
Assessment of differential efficacy according osteopathic practitioner profile (age/experience, perinatal specialization…) | at 10 days of life
Description of osteopathic dysfunctions frequencies diagnosed by osteopath. | at 10 days of life
Safety assessment measured by per-treatment DAN score | at 10 days of life
Curative efficacy of osteopathic treatment on nipple cracks, measured by the number of nipple cracks | at one month of life

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Baptiste MULLER, Doctor, Principal Investigator — Centre Hospitalier Universitaire de Nantes, France
Locations (1):
- Centre Hospitalier Universitaire de Nantes - Hôpital Mère-Enfant, Nantes, France

REFERENCES:
- [Derived] Danielo Jouhier M, Boscher C, Roze JC, Cailleau N, Chaligne F, Legrand A, Flamant C, Muller JB; NEOSTEO osteopath study group. Osteopathic manipulative treatment to improve exclusive breast feeding at 1 month. Arch Dis Child Fetal Neonatal Ed. 2021 Nov;106(6):591-595. doi: 10.1136/archdischild-2020-319219. Epub 2021 Mar 31. PMID 33789971